CLINICAL TRIAL: NCT05873192
Title: Presurgical Phase II Study of Talazoparib in Combination With Enzalutamide in de Novo Metastatic to Lymph Nodes Prostate Cancer
Brief Title: Presurgical Phase II Study of Talazoparib in Combination With Enzalutamide in Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0339; NCI-2023-03938 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; talazoparib; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADT plus Enzalutamide plus Talazoparib (Experimental): Participant will recive ADT plus Enzalutamide for a total of 8 weeks. After about 8 weeks of ADT and Enzalutamide treatment, participant will begin taking Talazoparib
  Interventions: Drug: ADT; Drug: Enzalutamide; Drug: Talazoparib; Drug: Degarelix; Drug: Luprolide

INTERVENTIONS:
Drug: ADT — Given by PO
  Other Names: Hormone Therapy
Drug: Enzalutamide — Given by PO
  Other Names: MDV3100; XTANDI®
Drug: Talazoparib — Given by PO
  Other Names: BMN 673; Talazoparib tosylate
Drug: Degarelix — Given PO or given INJ
Drug: Luprolide — Given PO or given INJ

SUMMARY:
To learn about the effectiveness of adding talazoparib to the standard of care treatment combination of androgen ablation therapy (hormone therapy, also known as ADT) and enzalutamide in patients with prostate cancer that has spread into the lymph nodes.

DETAILED DESCRIPTION:
Primary Objective:

•To evaluate the antitumor activity of presurgical talazoparib (PF-06944076) in combination with enzalutamide and androgen deprivation therapy (ADT) followed by surgery, in patients newly diagnosed with prostate cancer metastatic to lymph nodes (TxN1M0, TxNxM1a), as determined by the proportion of patients with undetectable prostate-specific antigen (PSA) 1 year after surgery.

Secondary Objectives:

* Analyze pathologic response in the primary tumor and metastatic lymph nodes to talazoparib in combination with enzalutamide and ADT in this population.
* Analyze 5-year disease-free survival and 5-year metastasis-free survival after talazoparib in combination with enzalutamide and ADT followed by surgical consolidation in this population.
* Evaluate the safety and tolerability of presurgical talazoparib in combination with enzalutamide and ADT in this population.
* Evaluate induction of a conditional homologous recombination deficient (HRD) state after 2 mos. of ADT and enzalutamide treatment relative to clinical and pathological outcomes.

Exploratory Objectives:

* To evaluate predictive and/or prognostic genomic and transcriptomic biomarkers associated with response to treatment or disease progression.
* To correlate data on intra-patient genomic heterogeneity from tumor biopsies and data from functional imaging with clinical benefit endpoints.
* To study possible mechanisms of resistance to study treatments through the comparative analysis of candidate biomarkers from paired pre-treatment, on therapy, and post-therapy tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with adenocarcinoma of the prostate that in the opinion of the urologist could be resected after response to systemic therapy. Ductal adenocarcinoma is permitted.
2. Patients must be regarded as acceptable surgical risk and confirm their intention to undergo radical prostatectomy at the end of the pre-surgical therapy.
3. ECOG performance status 2 or better.
4. All patients must have tumor staging and meet at least one of the following criteria:

   1. Either lymph node biopsy or lymph node dissection demonstrating lymph node metastasis by prostate cancer.
   2. Non-bulky (<5 cm) regional pelvic or distant lymphadenopathy visualized on CT/MRI/PET scan. Lymph node biopsy confirmation will be required if <2.0 cm or in atypical distribution*.
   3. The 2018 AJCC staging system will be followed.
5. Prior hormonal therapy (LHRH agonist/antagonist with or without first-generation antiandrogen) up to 6 weeks is permitted, provided any tumor biopsy specimen collected prior to initiation of ADT is made available for biomarker studies. If patient was started on first-generation antiandrogens, these would be discontinued prior to randomization.
6. Patients must agree to tissue collection for correlative studies at the specified timepoints. At the study entry, any previously collected diagnostic tumor biopsy blocks from primary and/or metastatic tissues must be provided.
7. Patients must have adequate bone marrow function defined as hemoglobin ³10 g/dL, an absolute peripheral neutrophil count (ANC) of ≥1,500/mm3 and platelet count of ≥100,000/mm3; no features suggestive of MDS/AML on peripheral blood smear; adequate hepatic function defined with a total bilirubin of ≤1.5 x upper limit of normal (ULN) (≤3 × ULN in subjects with Gilbert's disease), and AST/ALT ≤2.5 x ULN; adequate renal function defined as creatinine <1.5 x ULN or creatinine clearance ≥30 mL/min (measured or calculated with the Cockcroft-Gault Equation).
8. Medications known to lower the seizure threshold must be discontinued or substituted at least 4 weeks prior to study entry.
9. Patients or their partners must be surgically sterile or must agree to use one highly method or two effective methods of contraception while receiving study treatments and for at least 4 months thereafter. The definition of effective contraception should be in agreement with local regulation and based on the judgment of the principal investigator or a designated associate.
10. Patients must sign the current IRB approved informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution, and willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
11. All patients must have a surgical and medical oncology consult prior to signing informed consent.

Exclusion Criteria:

1. Patients with biopsy-proven small cell or sarcomatoid histology.
2. Patients with clinical or radiological evidence of bone or other extranodal metastasis.
3. Patients who have had prior chemotherapy, experimental agents for prostate cancer, or patients receiving >4 weeks of prior ADT will be excluded.
4. Treatment with estrogens, cyproterone acetate or glucocorticoids (at a dose >10 mg/day of prednisone equivalent) in the 4 weeks prior to scheduled Day 1 of treatment.
5. Gastrointestinal abnormalities such as inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection; active gastrointestinal bleeding as evidenced by hematemesis, hematochezia, or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy; malabsorption syndromes.
6. History or current diagnosis of MDS/AML, and/or history of any malignancy [other than the one treated in this study] which has a ≥ 30% probability of recurrence within 24 months (except for adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix or Ta urothelial carcinoma).
7. Known hypersensitivity to recombinant proteins, or any excipient contained in the drug formulation for talazoparib and/or enzalutamide.
8. Congenital long QT syndrome or Electrocardiogram (ECG) at screening with QT interval corrected using Fridericia's formula (QTcF) > 500 milliseconds.
9. Patients with any infectious process that, in the opinion of the investigator, could worsen or its outcome be affected as a result of the investigational therapy.
10. Patients with active or symptomatic viral hepatitis or chronic liver disease.
11. Patients with active pneumonitis or extensive bilateral lung disease of non-malignant etiology.
12. Patients with seizures or known condition that may pre-dispose to seizures (e.g., prior stroke or transient ischemic attack within 1 year to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy).
13. Patients with symptomatic congestive heart failure, unstable angina or myocardial infarction, coronary/peripheral artery bypass graft or repair, clinically significant ventricular arrhythmias, deep vein thrombosis or pulmonary embolism in the 6 months prior to randomization.
14. Persistently uncontrolled diabetes mellitus or HIV infection.
15. Inadequately controlled hypertension (defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >95 mmHg) despite antihypertensive medication, or prior history of hypertensive encephalopathy.
16. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
17. Anticipation of need for major surgical procedure during the course of the study other than as outlined by the protocol.
18. History of abdominal fistula or gastrointestinal perforation within 6 months prior to randomization.
19. Overt psychosis, mental disability, otherwise incompetent to give informed consent, or history of non-compliance.
20. Planned participation in any other experimental drug study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Amado Zurita-Saavedra, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org